CLINICAL TRIAL: NCT06035146
Title: Protective Ventilation in Patients With Lung Impairment on Mechanical Ventilation Controlled by the Mechanical Energy of the Respiratory System
Brief Title: Mechanical Ventilation in Patients With Lung Impairment Controlled by the Mechanical Energy of the Respiratory System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25/RVO-FNOs/2022
Record Dates: First submitted 2023-02-15; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: ARDS; Lung Injury, Ventilator Induced
Keywords: mechanical ventilation; adult respiratory distress syndrome; ventilator-induced lung injury; mechanical energy
MeSH Terms: conditions — Ventilator-Induced Lung Injury; Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: The study subjects will be randomized into two parallel groups.
Masking Description: No masking will be used in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mechanical energy monitoring (Experimental): In the study subjects randomized into this arm, the value of mechanical energy will be monitored during mechanical ventilation.
  Interventions: Procedure: Mechanical energy monitoring
- Conventional mechanical ventilation (Active Comparator): Study subjects randomized into this arm will receive conventional mechanical ventilation, to the best of the physician's knowledge.
  Interventions: Procedure: Conventional mechanical ventilation

INTERVENTIONS:
Procedure: Mechanical energy monitoring — Monitoring of the mechanical energy acting on the lung parenchyma during mechanical ventilation.
  Arms: Mechanical energy monitoring
Procedure: Conventional mechanical ventilation — The conventional procedure of mechanical ventilation controlled according to the physician's decision.
  Arms: Conventional mechanical ventilation

SUMMARY:
A project aimed at expanding the monitoring of mechanical energy (ME) in patients on mechanical ventilation (MV), with the aim of contributing to reducing the influence of the device for mechanical ventilation of patients on the lung parenchyma by setting parameters that will lead to lower ventilation energy.

According to the parameters set on the device for mechanical ventilation, the mechanical energy will be calculated, which the physician in the interventional arm of the study will be able to use to change the mechanical ventilation settings. The physician will follow the best clinical practice, and in the non-intervention group, the MV setting will be conventional.

DETAILED DESCRIPTION:
Mechanical ventilation (MV) in patients with acute respiratory failure (ARF) is one of the most common causes of hospitalization in the intensive care unit (ICU). ARF can be associated with severe forms of lung injury, the so-called ARDS (adult respiratory distress syndrome). Despite progress in the management of patients with ARDS, the mortality of these patients remains high, with in-hospital mortality reaching up to 45%. In patients with severe ARDS, mechanical ventilation can damage the lung parenchyma and cause ventilator-induced lung injury (VILI), which further worsens the patient's prognosis.

The result of setting the individual parameters of mechanical ventilation is the energy that the device exerts on the lung parenchyma, which ensures the opening of the lungs and a change in their volume related to gas exchange during breathing.

Routine laboratory values of blood gases and parameters of inflammation (CRP, PCT) will be recorded; which is part of routine clinical practice and standard patient care unrelated to the study.

As part of a prospective randomized study, a system for monitoring mechanical energy at the patient's bedside will be developed. Patients will be randomized into two groups - the intervention arm (mechanical ventilation controlled according to ME) and the non-intervention arm (conventional method of conducting mechanical ventilation).

ELIGIBILITY:
Inclusion Criteria:

* patients with fully controlled mechanical ventilation
* patients older than 18 years
* patients with lung disease (pneumonia, ARDS)
* expected duration of mechanical ventilation longer than 48 hours

Exclusion Criteria:

* pregnant women, when this fact is stated in the admission protocol
* inclusion in the study in a period longer than 24 hours from the start of mechanical ventilation (from admission to the Anesthesiology and Resuscitation Department)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The level of mechanical energy (in Joules/min) | up to 14 days
  The level of mechanical energy will be measured (in Joules/min) in both study arms.

SECONDARY OUTCOMES:
The number of days on mechanical ventilation | up to 14 days
  The number of days on mechanical ventilation will be observed in both study arms.
The effect of mechanical energy on patient mortality | up to 14 days
  The effect of mechanical energy on patient mortality will be analysed in both study arms. A mortality rate is the number of deaths due to a disease divided by the total population.
The effect of mechanical energy on hospital mortality | up to 8 weeks
  The effect of mechanical energy on hospital mortality will be analysed in both study arms. A mortality rate is the number of deaths due to a disease divided by the total population.

CONTACTS AND LOCATIONS:
Overall Officials: Filip Burša, MD,PhD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers. The data may be provided upon request.

REFERENCES:
- [Background] Papazian L, Calfee CS, Chiumello D, Luyt CE, Meyer NJ, Sekiguchi H, Matthay MA, Meduri GU. Diagnostic workup for ARDS patients. Intensive Care Med. 2016 May;42(5):674-685. doi: 10.1007/s00134-016-4324-5. Epub 2016 Mar 23. PMID 27007111
- [Background] Maca J, Jor O, Holub M, Sklienka P, Bursa F, Burda M, Janout V, Sevcik P. Past and Present ARDS Mortality Rates: A Systematic Review. Respir Care. 2017 Jan;62(1):113-122. doi: 10.4187/respcare.04716. Epub 2016 Nov 1. PMID 27803355
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Background] Rittayamai N, Brochard L. Recent advances in mechanical ventilation in patients with acute respiratory distress syndrome. Eur Respir Rev. 2015 Mar;24(135):132-40. doi: 10.1183/09059180.00012414. PMID 25726563
- [Background] Guerin C, Papazian L, Reignier J, Ayzac L, Loundou A, Forel JM; investigators of the Acurasys and Proseva trials. Effect of driving pressure on mortality in ARDS patients during lung protective mechanical ventilation in two randomized controlled trials. Crit Care. 2016 Nov 29;20(1):384. doi: 10.1186/s13054-016-1556-2. PMID 27894328
- [Background] Gattinoni L, Marini JJ, Pesenti A, Quintel M, Mancebo J, Brochard L. The "baby lung" became an adult. Intensive Care Med. 2016 May;42(5):663-673. doi: 10.1007/s00134-015-4200-8. Epub 2016 Jan 18. PMID 26781952
- [Background] de Prost N, Ricard JD, Saumon G, Dreyfuss D. Ventilator-induced lung injury: historical perspectives and clinical implications. Ann Intensive Care. 2011 Jul 23;1(1):28. doi: 10.1186/2110-5820-1-28. PMID 21906379
- [Background] Nieman GF, Satalin J, Andrews P, Habashi NM, Gatto LA. Lung stress, strain, and energy load: engineering concepts to understand the mechanism of ventilator-induced lung injury (VILI). Intensive Care Med Exp. 2016 Dec;4(1):16. doi: 10.1186/s40635-016-0090-5. Epub 2016 Jun 18. PMID 27316442
- [Background] Gattinoni L, Tonetti T, Cressoni M, Cadringher P, Herrmann P, Moerer O, Protti A, Gotti M, Chiurazzi C, Carlesso E, Chiumello D, Quintel M. Ventilator-related causes of lung injury: the mechanical power. Intensive Care Med. 2016 Oct;42(10):1567-1575. doi: 10.1007/s00134-016-4505-2. Epub 2016 Sep 12. PMID 27620287
- [Background] Cressoni M, Gotti M, Chiurazzi C, Massari D, Algieri I, Amini M, Cammaroto A, Brioni M, Montaruli C, Nikolla K, Guanziroli M, Dondossola D, Gatti S, Valerio V, Vergani GL, Pugni P, Cadringher P, Gagliano N, Gattinoni L. Mechanical Power and Development of Ventilator-induced Lung Injury. Anesthesiology. 2016 May;124(5):1100-8. doi: 10.1097/ALN.0000000000001056. PMID 26872367
- [Background] Chiumello D, Gotti M, Guanziroli M, Formenti P, Umbrello M, Pasticci I, Mistraletti G, Busana M. Bedside calculation of mechanical power during volume- and pressure-controlled mechanical ventilation. Crit Care. 2020 Jul 11;24(1):417. doi: 10.1186/s13054-020-03116-w. PMID 32653011
- [Background] Giosa L, Busana M, Pasticci I, Bonifazi M, Macri MM, Romitti F, Vassalli F, Chiumello D, Quintel M, Marini JJ, Gattinoni L. Mechanical power at a glance: a simple surrogate for volume-controlled ventilation. Intensive Care Med Exp. 2019 Nov 27;7(1):61. doi: 10.1186/s40635-019-0276-8. PMID 31773328
- [Background] Becher T, van der Staay M, Schadler D, Frerichs I, Weiler N. Calculation of mechanical power for pressure-controlled ventilation. Intensive Care Med. 2019 Sep;45(9):1321-1323. doi: 10.1007/s00134-019-05636-8. Epub 2019 May 17. No abstract available. PMID 31101961
- [Background] Serpa Neto A, Deliberato RO, Johnson AEW, Bos LD, Amorim P, Pereira SM, Cazati DC, Cordioli RL, Correa TD, Pollard TJ, Schettino GPP, Timenetsky KT, Celi LA, Pelosi P, Gama de Abreu M, Schultz MJ; PROVE Network Investigators. Mechanical power of ventilation is associated with mortality in critically ill patients: an analysis of patients in two observational cohorts. Intensive Care Med. 2018 Nov;44(11):1914-1922. doi: 10.1007/s00134-018-5375-6. Epub 2018 Oct 5. PMID 30291378
- [Background] Mietto C, Malbrain ML, Chiumello D. Transpulmonary pressure monitoring during mechanical ventilation: a bench-to-bedside review. Anaesthesiol Intensive Ther. 2015;47 Spec No:s27-37. doi: 10.5603/AIT.a2015.0065. Epub 2015 Nov 17. PMID 26575165
- [Derived] Bursa F, Frelich M, Sklienka P, Kucerova Z, Sagan J, Oczka D, Penhaker M, Burda M, Maca J. Protective mechanical ventilation controlled by the real-time mechanical power measurement. J Clin Monit Comput. 2025 Oct 11. doi: 10.1007/s10877-025-01369-w. Online ahead of print. PMID 41075121